CLINICAL TRIAL: NCT01802424
Title: The FRIENDS-program as Indicative Prevention for Children and Adolescents With Symptoms of Anxiety and Depression
Brief Title: FRIENDS as an Indicative Prevention Program in Norway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 71 FRIENDS
Record Dates: First submitted 2013-02-21; First posted 2013-03-01 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Anxiety
Keywords: Open trial; Indicative prevention; Youth anxiety; Cognitive behavioral therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The Friends program (Experimental): Youth with increased levels of anxiety are thought to regulate their fear by recognizing bodily cues, learning relaxation, regulating thoughts and feelings and expose themselves to situations and objects that activate their anxiety.
  Interventions: Behavioral: The Friends program

INTERVENTIONS:
Behavioral: The Friends program — The Friends program is a ten weeks group interventions based on principles from Cognitive Behavioural Therapy aimed at ameliorating symptoms of anxiety and depression in children and adolescents. There are age-specific versions of the manual, one for children 8-12 years and one for adolescents 12-15 years.

SUMMARY:
The purpose of this pilot-study is to evaluate a cognitive behavioral program, the Friends-program, as indicated prevention for anxious youth. The youths are recruited by school nurses who will also lead the intervention groups applying the Friends-manual.

ELIGIBILITY:
Inclusion Criteria:

* subclinical to clinical symptoms of anxiety with or without comorbid symptoms of depression

Exclusion Criteria:

* previously diagnosed with conduct disorder, major life-crises that needs to be attended to, serious school refusal, Obsessive Compulsive Disorder, mental retardation or autism.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in anxiety symptoms from baseline to 12 months after completing the FRIENDS program, measured by the Spence Children Anxiety Scale (SCAS) | When completing the intervention and 3months and 12 months after having completed the intervention

SECONDARY OUTCOMES:
Changes in life-quality (measured by KINDL)from baseline to 12 months after completing the FRIENDS program | When completing the intervention and 3months and 12 months after having completed the intervention
Changes in depressive symptoms (measured by the Short Mood and Feeling questionnaire)from baseline to 12 months after completing the FRIENDS program | When completing the intervention and 3months and 12 months after having completed the intervention
Changes in psychosocial functioning (measured by the Strengths and difficulties questionnaire)from baseline until 12 months after having completed the FRIENDS program | When completing the intervention and 3months and 12 months after having completed the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bente SM Haugland, PhD, Principal Investigator — Uni Research Health
Locations (1):
- Fjell municipality, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No